CLINICAL TRIAL: NCT05456685
Title: Multicenter, Open-label, Phase 2 Study of Carboplatin Plus Mirvetuximab Soravtansine Followed by Mirvetuximab Soravtansine Continuation in FRα Positive, Recurrent Platinum-sensitive, High-grade Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancers Following 1 Prior Line of Platinum-based Chemotherapy
Brief Title: Mirvetuximab Soravtansine (MIRV) With Carboplatin in Second-line Treatment of Folate Receptor Alpha (FRα) Expressing, Platinum-sensitive Epithelial Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMGN853-0420; 2022-501220-14-00 (Other: EU CT)
Record Dates: First submitted 2022-06-29; First posted 2022-07-13 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: High Grade Ovarian Cancer; Primary Peritoneal Cancer; Fallopian Tube Cancer
Keywords: platinum sensitive; folate-receptor alpha expression; antibody-drug conjugate; cancer; ovarian neoplasm; high-grade ovarian
MeSH Terms: conditions — Fallopian Tube Neoplasms; Neoplasms; Ovarian Neoplasms | interventions — mirvetuximab soravtansine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- MIRV + Carboplatin (Experimental): On Day 1 of every 3-week cycle (Q3W) for 6 cycles, MIRV will be given at the dosage of 6 mg/kg of AIBW along with carboplatin given at area under the AUC5 administered through intravenous (IV) infusion (maximum dosing per National Comprehensive Cancer Network [NCCN] guidelines [NCCN 2021]). Upon completion of carboplatin plus MIRV treatment, single-agent MIRV will be continued at the tolerated dose on Day 1 Q3W in participants with investigator determined stable disease (SD), complete response (CR) or partial response (PR).
  Interventions: Drug: Mirvetuximab soravtansine; Drug: Carboplatin

INTERVENTIONS:
Drug: Mirvetuximab soravtansine — Mirvetuximab Soravtansine (MIRV) is an investigational antibody drug conjugate designed to selectively kill cancer cells. The antibody (protein) part of MIRV targets tumors by delivering a cell-killing drug to the tumor cells carrying a tumor-associated protein called FRα. It is being developed for the treatment of participants with recurrent platinum-sensitive, high grade epithelial ovarian, primary peritoneal, or fallopian tube cancers with FRα expression. FRα positivity will be defined by the Ventana FOLR1 Assay.
  Other Names: MIRV; IGN853
Drug: Carboplatin — Carboplatin is considered to be the treatment agent of choice in relapsed PSOC.

SUMMARY:
IMGN853-0420 is a multicenter, open-label, phase 2 study of carboplatin plus mirvetuximab soravtansine followed by mirvetuximab soravtansine continuation in folate receptor-alpha positive, recurrent platinum sensitive, high-grade epithelial ovarian, primary peritoneal, or fallopian tube cancer following 1 prior line of platinum-based chemotherapy.

DETAILED DESCRIPTION:
This Phase 2 study is designed to evaluate the efficacy and safety of MIRV in combination with carboplatin followed by MIRV continuation in FRα-positive participants with recurrent platinum-sensitive ovarian cancer (PSOC) following 1 prior line of platinum-based chemotherapy. Upon completion of carboplatin plus MIRV combination chemotherapy (6 cycles), participants without progressive disease will continue on single-agent MIRV. Participants must have confirmation of FRα positivity by the Ventana folate receptor 1 (FOLR1) Assay.

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥ 18 years of age.
2. Must have an Eastern Cooperative Oncology Group Performance Status of 0 or 1.
3. Must have a confirmed diagnosis of high-grade serous epithelial ovarian, primary peritoneal, or fallopian tube cancer.
4. Must have relapsed after 1 prior line of platinum-based chemotherapy.
5. Must have platinum-sensitive disease defined as radiographic progression greater than 6 months from last dose of platinum-based chemotherapy. Note: Progression should be calculated from the date of the last administered dose of platinum therapy to the date of the radiographic imaging showing progression.
6. If available locally and is the standard of care, breast cancer susceptibility gene (BRCA) testing on the tumor or prior germline testing is required for eligibility, and will need to be done prior to study entry. Somatic and germline BRCA-positive participants must have received prior treatment with a poly adenosine phosphate-ribose polymerase inhibitor (PARPi) unless documented as clinically contraindicated.
7. Must have at least 1 lesion that meets the definition of measurable disease by RECIST v1.1 (radiologically measured by the investigator).
8. Must provide an archival tumor tissue block or slides, or undergo procedure to obtain a new biopsy using a low-risk, medically routine procedure for immunohistochemistry (IHC) confirmation of FRα positivity; FRα-expressing tumors will be defined and classified by the Ventana FOLR1 Assay into low, medium, and high expressions defined as 25%-49%, 50%-74%, and ≥ 75% of tumor cells with PS2+ staining intensity, respectively. Must have confirmation of FRα positivity of ≥ 25% of tumor staining at ≥ 2+ intensity for entry into the study.
9. Must have stabilized or recovered (Grade 1 or baseline) from all prior therapy-related toxicities (except alopecia) and have discontinued any maintenance therapy at least 4 weeks before the first dose of carboplatin plus MIRV.
10. Must have completed any major surgery at least 4 weeks before the first dose of carboplatin plus MIRV and have recovered or stabilized from the side effects of prior surgery before the first dose of carboplatin plus MIRV.
11. Must have adequate hematologic, liver, and kidney functions defined as:

    1. Absolute neutrophil count ≥ 1.5 × 10^9/ liter(L) (1500/ microliter [μL]) without granulocyte colony-stimulating factor or long-acting white blood cell growth factors in the 10 days prior to the Cycle 1 Day 1 (C1D1) dose
    2. Platelet count ≥ 100 × 109/L (100,000/μL) without platelet transfusion in the 10 days prior to the C1D1 dose
    3. Hemoglobin ≥ 9.0 grams/deciliter (g/dL) without packed red blood cell transfusion in the 14 days prior to the C1D1 dose
    4. Serum creatinine ≤ 1.5 × upper limit of normal (ULN)
    5. Aspartate aminotransferase and alanine aminotransferase ≤ 3.0 × ULN
    6. Serum bilirubin ≤ 1.5 × ULN (participants with documented diagnosis of Gilbert syndrome are eligible if total bilirubin < 3.0 × ULN)
    7. Serum albumin ≥ 2 g/dL
12. Must be willing and able to sign the informed consent form (ICF) and to adhere to the protocol requirements.
13. Females of childbearing potential (FCBP) must agree to use highly effective contraceptive method(s) while on study medication and for at least 3 months after the last dose of MIRV and 6 months after the last dose of carboplatin.
14. FCBP must have a negative pregnancy test within the 4 days prior to the C1D1 dose.

Exclusion Criteria:

1. Participants with endometrioid, clear cell, mucinous, or sarcomatous histology, mixed tumors containing any of the above types, or low-grade/ borderline ovarian tumor
2. More than one line of prior chemotherapy. Lines of prior anticancer therapy are counted with the following considerations:

   1. Neoadjuvant ± adjuvant therapies are considered 1 line of therapy if the neoadjuvant and adjuvant correspond to 1 fully predefined regimen; otherwise, they are counted as 2 prior regimens.
   2. Maintenance therapy (eg, bevacizumab, PARPi) will be considered part of the preceding line of therapy (ie, not counted independently).
3. Participants with prior wide-field radiotherapy affecting at least 20% of the bone marrow
4. Participants with > Grade 1 peripheral neuropathy per Common Terminology Criteria for Adverse Events (CTCAE)
5. Participants with active or chronic corneal disorders, history of corneal transplantation, or active ocular conditions requiring ongoing treatment/ monitoring, such as uncontrolled glaucoma, wet age-related macular degeneration requiring intravitreal injections, active diabetic retinopathy with macular edema, macular degeneration, presence of papilledema, or monocular vision
6. Participants with serious concurrent illness or clinically relevant active infection, including, but not limited to the following:

   1. Active hepatitis B virus (HBV) or hepatitis C virus (HCV)or C infection (whether or not on active antiviral therapy)
   2. HIV infection if inclusion clarifying eligibility for HIV positive participants is not met
   3. Active cytomegalovirus infection
   4. Any other concurrent infectious disease requiring IV antibiotics within 2 weeks prior to the first dose of carboplatin plus MIRV Note: Testing at screening is not required for the above infections unless clinically indicated.
7. Participants with a history of multiple sclerosis or other demyelinating disease and/or Lambert-Eaton syndrome (paraneoplastic syndrome)
8. Participants with clinically significant cardiac disease including, but not limited to, any of the following:

   1. Myocardial infarction ≤ 6 months prior to first dose
   2. Unstable angina pectoris
   3. Uncontrolled congestive heart failure (New York Heart Association > class II)
   4. Uncontrolled ≥ Grade 3 hypertension (per CTCAE)
   5. Uncontrolled cardiac arrhythmias
9. Participants with a history of hemorrhagic or ischemic stroke within 6 months prior to enrollment
10. Participants with a history of cirrhotic liver disease (Child-Pugh Class B or C)
11. Participants with a previous clinical diagnosis of noninfectious interstitial lung disease, including noninfectious pneumonitis (exception: Grade 1 noninfectious pneumonitis diagnosed on or within 6 weeks after treatment with an immunotherapeutic agent used in the treatment of their malignancy that has resolved per investigator or resolution of the radiologic findings)
12. Participants requiring use of folate-containing supplements (eg, folate deficiency)
13. Participants with prior hypersensitivity to monoclonal antibodies (mAb)
14. Females who are pregnant or breastfeeding
15. Participants who received prior treatment with MIRV or other FRαtargeting agents
16. Participants with untreated or symptomatic central nervous system metastases
17. Participants with a history of other malignancy within 3 years before enrollment Note: Participants with tumors with a negligible risk for metastasis or death (eg, adequately controlled basal-cell carcinoma or squamous-cell carcinoma of the skin, or carcinoma in situ of the cervix or breast) are eligible.
18. Prior known hypersensitivity reactions or known contraindications to study drugs or any of their excipients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to 3 years
  ORR following carboplatin plus MIRV combination as measured by the investigator and assessed according to RECIST v1.1, defined as the proportion of confirmed responders (CR or PR) among participants with FRα expression of ≥ 50%
  o ORR following carboplatin plus MIRV combination will also be measured, as a sensitivity analysis, by a blinded independent central review (BICR) in the same participant population

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 3 years
  ORR, defined as the proportion of confirmed responders (CR or PR) following carboplatin plus MIRV combination, as measured by the investigator and assessed according to RECIST v1.1, among patients with FRα expression of ≥ 25% of tumor cells with PS2+ staining intensity who have measurable disease per RECIST v1.1 at inclusion.
  o ORR will also be measured by a BICR, as a sensitivity analysis, in the same patient population.
Duration of Response (DOR) | Up to 3 years
  DOR, defined as the time from first response to radiological progressive disease (PD) or death, whichever occurs first, following carboplatin plus MIRV followed by MIRV continuation by the investigator and assessed according to RECIST v1.1 among efficacy evaluable participants:
  * with FRα expression of ≥ 50% of tumor cells with PS2+ staining and
  * with FRα expression of ≥ 25% of tumor cells with PS2+ staining
  * DOR in the above populations will also be measured by BICR
Progression Free Survival (PFS) | Up to 3 years
  PFS as measured by the investigator and by BICR in participants with
  * FRα expression of ≥ 50% of tumor cells with PS2+ staining and
  * FRα expression of ≥ 25% of tumor cells with PS2+ staining
Overall Survival (OS) | Up to 3 years
  OS in participants with
  * FRα expression of ≥ 50% of tumor cells with PS2+ staining and
  * FRα of ≥ 25% of tumor cells with PS2+ staining
Cancer Antigen (CA)-125 Response | Up to 3 years
  CA-125 response as measured by the investigator, per Gynecologic Cancer Intergroup (GCIG), in the efficacy evaluable participants with
  * FRα expression of ≥ 50% of tumor cells with PS2+ staining and
  * FRα expression of ≥ 25% of tumor cells with PS2+ staining
Number of Participants With treatment Emergent Adverse Events (TEAEs) | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (69):
- United States (35):
  - University of Arizona Cancer Center /ID# 268906, Tucson, Arizona
  - Women'S Cancer Research Network - Cogi /ID# 268912, Fresno, California
  - Providence - St. Jude Medical /ID# 268911, Fullerton, California
  - Moores Cancer Center /ID# 268888, La Jolla, California
  - USC Norris Comprehensive Cancer Center /ID# 268964, Los Angeles, California
  - University of California Los Angeles Medical Center /ID# 268883, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian /ID# 268907, Newport Beach, California
  - UC Davis Comprehensive Cancer Center /ID# 269085, Sacramento, California
  - Scripps Md Anderson - Prebys Cancer Center /ID# 268966, San Diego, California
  - California Pacific Medical Center - Van Ness Campus /ID# 268886, San Francisco, California
  - Smilow Cancer Hospital at Yale New Haven /ID# 268889, New Haven, Connecticut
  - AdventHealth Orlando /ID# 268920, Orlando, Florida
  - Sarasota Memorial Hospital /ID# 268882, Sarasota, Florida
  - Moffitt Cancer Center /ID# 269089, Tampa, Florida
  - Winship Cancer Institute of Emory University /ID# 268913, Atlanta, Georgia
  - Northwestern University- Robert H. Lurie Comprehensive Cancer Center /ID# 268957, Chicago, Illinois
  - Women'S Cancer Care /ID# 268898, Covington, Louisiana
  - Massachusetts General Hospital /ID# 268879, Boston, Massachusetts
  - Dana-Farber Cancer Institute /ID# 268881, Boston, Massachusetts
  - Karmanos Cancer Institute - Detroit /ID# 268890, Detroit, Michigan
  - Washington University School of Medicine - St. Louis /ID# 268897, St Louis, Missouri
  - The Center Of Hope /ID# 268884, Reno, Nevada
  - Md Anderson Cancer Center At Cooper /ID# 268885, Camden, New Jersey
  - Holy Name Medical Center /ID# 268903, Teaneck, New Jersey
  - University of New Mexico Comprehensive Cancer Center /ID# 268961, Albuquerque, New Mexico
  - Presbyterian Rust Medical Center /ID# 278582, Rio Rancho, New Mexico
  - Long Island Jewish Medical Center /ID# 268909, New Hyde Park, New York
  - Columbia University Irving Medical Center /ID# 268887, New York, New York
  - University of North Carolina Medical Center /ID# 268963, Chapel Hill, North Carolina
  - Duke Cancer Center Macon Pond /ID# 268910, Raleigh, North Carolina
  - OU Health - Stephenson Cancer Center /ID# 268878, Oklahoma City, Oklahoma
  - Women & Infants Hospital /ID# 268895, Providence, Rhode Island
  - MUSC Hollings Cancer Center /ID# 268892, Charleston, South Carolina
  - University of Texas - Southwestern Medical Center /ID# 268891, Dallas, Texas
  - Duplicate_Kadlec Clinic Heme-Onc /ID# 268580, Kennewick, Washington
- Belgium (3):
  - Cliniques Universitaires UCL Saint-Luc /ID# 268916, Brussels, Brussels Capital
  - Universitair Ziekenhuis Leuven /ID# 268914, Leuven, Vlaams-Brabant
  - Duplicate_CHU de Liege /ID# 268918, Liège
- Canada (5):
  - BC Cancer - Vancouver /ID# 268901, Vancouver, British Columbia
  - Universite de Montreal - Hopital Maisonneuve-Rosemont /ID# 268902, Montreal, Quebec
  - Centre Hospitalier De L'Universite De Montreal - Hopital Saint-Luc /ID# 268899, Montreal, Quebec
  - McGill University Health Centre - Glen Site /ID# 269084, Montreal, Quebec
  - Centre Hospitalier Universite De Sherbrooke - Hôtel-Dieu Hospital /ID# 268900, Sherbrooke, Quebec
- Georgia (5):
  - American Hospital Tbilisi /ID# 268947, Tbilisi
  - High Technology Hospital MedCenter /ID# 268946, Tbilisi
  - Israeli-Georgian Medical Research Clinic Helsicore /ID# 268950, Tbilisi
  - Caraps Medline /ID# 268948, Tbilisi
  - Duplicate_Consilium Medulla Multiprofile Clinic /ID# 268951, Tbilisi
- Spain (13):
  - Complejo Hospitalario Universitario A Coruña /ID# 268930, A Coruña, A Coruna
  - Institut Català d'Oncologia (ICO) - Badalona /ID# 268929, Badalona, Barcelona
  - Hospital Universitario Reina Sofia /ID# 269657, Córdoba, Cordoba
  - Clinica Universidad de Navarra - Pamplona /ID# 268940, Pamplona, Navarre
  - Complejos Hospitalario Universitario de Badajoz /ID# 268937, Badajoz
  - Usp Instituto Universitario Dexeus /ID# 268931, Barcelona
  - Hospital Universitario Vall de Hebron /ID# 268926, Barcelona
  - Hospital Universitario Arnau de Vilanova de Lleida /ID# 268939, Lleida
  - Clinica Universidad de Navarra - Madrid /ID# 268935, Madrid
  - Hospital Universitario Fundación Jiménez Díaz /ID# 268938, Madrid
  - Hospital Universitario 12 de Octubre /ID# 268936, Madrid
  - Hospital Universitario HM Sanchinarro /ID# 268932, Madrid
  - Hospital Clínico Universitario de Valencia /ID# 268933, Valencia
- United Kingdom (8):
  - Hammersmith Hospital /ID# 268945, London, England
  - Guy's Hospital /ID# 269083, London, Greater London
  - The Royal Marsden - Chelsea /ID# 268943, London, Greater London
  - Mount Vernon Hospital /ID# 268942, Northwood, Greater London
  - Nottinghamshire Healthcare NHS Foundation Trust /ID# 269087, Nottingham, Nottinghamshire
  - Musgrove Park Hospital /ID# 269088, Taunton, Somerset
  - The Royal Marsden - Sutton /ID# 268941, Sutton, Surrey
  - The Christie /ID# 268944, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=IMGN853-0420